CLINICAL TRIAL: NCT03272919
Title: Chemotherapy Induced Peripheral Neuropathy (CIPN): A Pilot Study of Intraneural Facilitation for Managing Chemotherapy-Induced Peripheral Neuropathy
Brief Title: Chemotherapy Induced Peripheral Neuropathy (CIPN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Gayathri Nagaraj, Associate Professor of Medicine, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5170197
Record Dates: First submitted 2017-08-08; First posted 2017-09-06 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Breast Cancer, Peripheral neuropathy, Taxol, carboplatin
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Investigational INF (Experimental): Intraneural Facilitation (INF) treatment is an effective way to restore blood flow to damaged nerves as neuropathy is strongly impacted by reduced blood flow.
  Interventions: Other: Arm 1: Investigational INF
- Arm 2: Standardized muscle stretching and strengthen (Other): subjects will receive a standardized program of muscle stretching and strengthening exercise twice a week for six weeks under the supervision of treating physical therapist
  Interventions: Other: Arm 2: standardized muscle stretching and strength

INTERVENTIONS:
Other: Arm 1: Investigational INF — INF utilizes three holds or positions, which widens tiny openings in arteries surrounding nerves and improves blood flow to targeted nerves. The improved blood flow in these nerves stimulates healing and reduces or even stops nerve pain.
  Arms: Arm 1: Investigational INF
Other: Arm 2: standardized muscle stretching and strength — subjects will receive a standardized program of muscle stretching and strengthening exercise under the supervision of treating physical therapist.
  Arms: Arm 2: Standardized muscle stretching and strengthen

SUMMARY:
Chemotherapy induced peripheral neuropathy (CIPN) is a common side effect of many forms of chemotherapy having a negative impact on the quality of life for cancer survivors due to numbness, decreased sensation, pain (of various intensities in the extremities), gait/balance problems, and difficulty with fine motor skills of the hands and fingers.To date, there are no preventive modalities to mitigate CIPN development.When CIPN becomes intolerable, optimal doses of chemotherapy have to be reduced or discontinued, which may affect a patient's overall survival. Intraneural facilitation (INF) is a technique developed by physical therapists at Loma Linda University after careful study of the structure, pathophysiology and biomechanics of peripheral nerves. The focus of INF is restoration of circulation to an ischemic nerve. INF has been offered to subjects receiving treatment at LLUCC with anecdotal success. The purpose of this study is to evaluate INF as a treatment modality under the rigor of scientific inquiry to determine its effectiveness as a viable treatment option for breast cancer patients with CIPN.

DETAILED DESCRIPTION:
STUDY OUTLINE: This is a single institution study. Patients with newly diagnosed breast cancer stages I to III with any biomarker status (ER, PR and HER), without preexisting peripheral neuropathy planning to receive treatment with platinum-based compounds (Carboplatin and Cisplatin) and/or taxanes (Docetaxel and Paclitaxel) and chemotherapy naive patients with gynecologic cancers including ovarian, uterine, and cervical cancer planning to receive definitive number of platinum-based compounds (carboplatin or cisplatin) and/or taxanes (docetaxel and paclitaxel) chemotherapy are potential study patients.

Subjects will be randomized into one of two treatment arms within 3 weeks of starting the offending chemotherapy agents after fulfilling the other study eligibility requirements. Arm 1 (investigational) will receive INF twice a week for six weeks by the same treating physical therapist (physical therapist #1). Arm 2 (control) will receive a standardized program of muscle stretching and strengthening exercises twice a week for 6 weeks under the supervision of treating physical therapist #1. Actual treatment time for both modalities is approximately 45 minutes. Measurements used to detect the presence and degree of peripheral neuropathy will be administered by the same assessment physical therapist (physical therapist #2) at baseline and at the end of weeks 3, 6, and 3 months post last physical therapy treatment. Assessment tools are: ultrasound imaging on the popliteal and posterior tibia artery, the 20-item Pain Quality Assessment Scale (PQAS, specifically addresses neuropathological symptomatology), the National Comprehensive Cancer Network (NCCN) Distress thermometer (DT), and the Michigan Neuropathy Screening Instrument (MNSI) will be assessed and recorded along with treatment adherence. Treating physician will be recording National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) neuropathy score and performance status at routine intervals during and after chemotherapy.

Objectives

Primary objective

• To compare the degree of neuropathy and distress between Arm 1 receiving INF therapy compared to Arm 2 receiving usual care of muscle stretching and strengthening exercises based on standardized measurements (PQAS, MNSI, NCCN DT, and AE assessment).

Secondary objectives

* To compare the Ultrasound measurements of peak systolic velocity, volume flow and pulsatility of popliteal and posterior tibia artery between the two treatment arms for assessing differences in vascular perfusion.
* To compare the rate of any dose reductions and premature chemotherapy discontinuation rates due to peripheral neuropathy between Arm 1 receiving INF therapy compared to Arm 2 receiving standardized program of muscle stretching and strengthening exercises.
* To compare subject acceptability, burden and satisfaction with the assigned physical therapy modality between the two arms based on patient satisfaction questionnaire administered at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed stages I to III breast cancer patients with any biomarker status (ER, PR and HER) receiving treatment with platinum-based compounds (Carboplatin and Cisplatin) and/or taxanes (Docetaxel and Paclitaxel).
* Chemotherapy naive patients with gynecologic cancers including ovarian, uterine, and cervical cancer planning to receive definitive number of platinum-based compounds (carboplatin or cisplatin) and/or taxanes (docetaxel and paclitaxel) chemotherapy.
* Planned to receive a minimum of 4 cycles of treatment with either of the offending chemotherapy agents (a cycle of weekly paclitaxel is considered 3 doses).
* Women aged ≥ 18 years at signing of informed consent
* No pre-existing peripheral neuropathy (WPPN)
* ECOG status 0 or 1
* Able to provide written, informed consent to participate in the study and follow the study procedures.
* Cannot participate in another non-medical intervention/therapy for peripheral neuropathy
* Cannot receive more than 3 weeks of treatment with implicating chemotherapy prior to start of study assigned therapy.

Exclusion Criteria:

* Male
* Preexisting peripheral neuropathy.
* Previous exposure to any of the implicated chemotherapy agents within the last 5 years (platinum-based compounds, vinca alkaloids and/or taxanes) that could potentially cause peripheral neuropathy
* Evidence of significant medical illness, or psychiatric illness/social situation that would, in the investigator's judgment, make the patient inappropriate for this study.
* Stage IV or metastatic breast cancer
* Any physical or neurological disability that would preclude patients from participating in physical therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women aged ≥ 18 years at signing of informed consent
Enrollment: 44 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Descriptive Statistics to measure the degree of peripheral neuropathy in the two arms based on the PQAS score. | upto 3 months post completion of assigned treatment
  The 20 item PQAS measures self reported aspects of nociceptive and neuropathic pain (intensity, sensation, depth, location) on a scale of 0 to 10.
Descriptive Statistics to measure the degree of distress in the two arms based on NCCN- DT | upto 3 months post completion of assigned treatment
  Study participants self report distress based on National Comprehensive Cancer Network's Distress Thermometer (DT) measures distress on a scale of 0 = no distress, 10=extreme distress.
Descriptive Statistics to measure the degree of peripheral neuropathy in the two arms based on MSNI scores | upto 3 months post completion of assigned treatment
  The MSNI is a physical screening instrument of the lower legs and feet for the assessment of neuropathy using visual inspection, vibration sensation, ankle reflexes and monofilament testing producing a score of 0 being normal and 10 meaning significant neuropathy as measured by the assessing physical therapist
Descriptive Statistics to measure the degree of peripheral neuropathy in the two arms based on CTCAE grading | upto 3 months post completion of assigned treatment
  The CTCAE measures peripheral sensory neuropathy on a scale of 1=asymptomatic to 5=death as measured by the treating physician

SECONDARY OUTCOMES:
Measure the peak systolic velocity on ultrasound imaging in the popliteal and posterior tibia artery in the two arms. | upto 3 months post completion of assigned treatment
  Ultrasound imaging will be administered before and after treatment on the measurement days for subjects in both Arm 1 and Arm 2
Measure the rate of premature chemotherapy discontinuation due to peripheral neuropathy by treatment group | upto 3 months post completion of assigned treatment
  The completion and premature discontinuation rates due to peripheral neuropathy for each subject will be counted for each Arm.
Measure the rate of dose reductions in chemotherapy due to peripheral neuropathy by treatment group | upto 3 months post completion of assigned treatment
  The dose reductions in chemotherapy due to peripheral neuropathy for each subject will be measured for each Arm.
Questionnaire to survey patients on acceptability, satisfaction and burden of treatment | upto 3 months post completion of assigned treatment.
  A written survey of 10 questions regarding subject acceptance, burden and satisfaction will be administered to each subject in both Arms at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gayathri Nagaraj, MD, Principal Investigator — Loma Linda University Medical Center; Ellen D'Errico, PHD, Principal Investigator — Loma Linda University School of Nursing
Locations (1):
- Loma Linda Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No